CLINICAL TRIAL: NCT00686140
Title: Celecoxib as Add-on Therapy to Risperidone Versus Risperidone Alone in First-Episode and Drug-naive Patients With Schizophrenia
Brief Title: A Double-blind and Randomized Trial of Celecoxib Added to Risperidone in Treatment-naive First-episode Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Director, Biological Psychiatry Center, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03T-459; SCH-A01; SMRI 03T-459 (Other Grant/Funding Number: SMRI 03T-459)
Record Dates: First submitted 2006-06-10; First posted 2008-05-29 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; clinical trial; risperidone; immune; celecoxib
MeSH Terms: conditions — Schizophrenia | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celecoxib, immune adjustor (Experimental): Celecoxib
  Interventions: Drug: celecoxib
- Placebo (Placebo Comparator): Placebo looks like the active drug celecoxib, with the same dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: celecoxib — 400mg/day, twice a day, 12 weeks
  Other Names: Celebrex(R)
  Arms: Celecoxib, immune adjustor
Drug: Placebo — twice a day, 12 weeks
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled trial of celecoxib as an add-on therapy to risperidone compared to risperidone plus placebo in the treatment of 200 treatment-naive first-episode patients with schizophrenia. The study addresses an immune dysfunction hypothesis of schizophrenia.

DETAILED DESCRIPTION:
OBJECTIVE: Evidences of high levels of activating cytokines in the CSF and signs of CNS inflammation have suggested that an inflammatory/immunological pathogenesis may exist in a subgroup of schizophrenic patients. We hypothesize that anti-inflammatory therapy by using an add-on agent together with a well-proven neuroleptic may have favorable effects on some schizophrenic patients.

METHODS:

1. Clinical Trial: This is a randomized, double-blind and parallel controlled trial in treatment-naive first-episode patients with schizophrenia. The study consists of a 1-week stabilization phase, followed by 12 weeks of double-blind treatment. The total trial duration is 13 weeks.
2. Assessment Procedures:

2.1. Primary Outcome Variable-psychopathology: Assessment instruments include the Positive and Negative Syndrome Scale (PANSS) (Kay et al, 1987), the Assessment of Negative Symptoms (SANS) (Andreasen 1981) and the Clinical Global Impression (ICG). Patients are interviewed at screening, at week-4, at week-1, at baseline and at every two weeks, for a total of 12 ratings.

2.2. Cognitive tests: A comprehensive battery of tests encompassing the cognitive domains of executive function, attention, memory, perception, and general intellect is administered twice at baseline and at the end of 16-week treatment by a trained psychologist. Scoring follows standardized procedures. The Wisconsin Card Sorting Test (WCST) (Heaton et al, 1993) is administered as a measure of executive function. The N-back (0-3 back) test is administered as a measure of working memory. Logical Memory I and II, Verbal Paired Associates I and II, Visual Reproduction I and II and Digits Forward from the Wechsler Memory Scale-Revised (WMS-R) (Wechsler, 1987) are administered as a tests of episodic memory. The Distractibility version of Gordon Continuous Performance Test (CPT)is administered as a test of attention. A four-subtest version of the Wechsler Adult Intelligence Scale-Revised (WAIS-R), (Wechsler, 1981; Missar et al, 1994) consisting of the Arithmetic, Similarities, Picture Completion, and Digit Symbol Substitution tests is administered to obtain an estimate of current Full-Scale Intelligence Quotient (FSIQ).

2.3. Side Effects: Parkinsonism is rated with the Simpson-Angus Scale for extrapyramidal side effects (SAS, Simpson and Angus, 1970). The Abnormal Involuntary Movement Scale (AIMS) (Guy, 1978) is chosen to assess tardive dyskinesia (TD) severity. All of the AIMS and Simpson-Angus Rating Scales are administered by the same investigator, at screening, at week-4, at week-1, at baseline and at baseline and at every two weeks, for a total of 12 ratings.

2.4.Serum Measures: IL-2, IL-6, IL-8 and IL-10 concentrations

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizophreniform disorder;
* Duration of symptoms not longer than 60 months;
* No prior treatment with antipsychotic medication or, if previously treated, a total lifetime usage of less than 14 days;
* Between 16 and 40 years of age; and
* Current psychotic symptoms of moderate severity.

Exclusion Criteria:

* A DSM-IV Axis I diagnosis other than schizophrenia or schizophreniform;
* Documented disease of the central nervous system that can interfere with the trial assessments including, but not limited to stroke, tumor, Parkinson's disease, Huntington's disease, seizure disorder, history of brain trauma resulting in significant impairment, chronic, infection;
* Acute, unstable and/or significant and untreated medical illness (e.g., infection, unstable diabetes, uncontrolled hypertension);
* A clinically significant ECG abnormality in the opinion of the investigator;
* Pregnant or breast-feeding female;
* Use of disallowed concomitant therapy;
* History of severe allergy or hypersensitivity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
PANSS | 12 weeks

SECONDARY OUTCOMES:
CGI | 12 weeks
AIMS | 12 weeks
Cognition | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lian Y Cao, M.D., Study Chair — Beijing HuiLongGuan Hospital
Locations (1):
- Beijing HuiLongGuan Hospital, Beijing, China

REFERENCES:
- [Derived] Wang DM, Chen DC, Xiu MH, Wang L, Kosten TR, Zhang XY. A double-blind, randomized controlled study of the effects of celecoxib on clinical symptoms and cognitive impairment in patients with drug-naive first episode schizophrenia: pharmacogenetic impact of cyclooxygenase-2 functional polymorphisms. Neuropsychopharmacology. 2024 Apr;49(5):893-902. doi: 10.1038/s41386-023-01760-8. Epub 2023 Oct 30. PMID 37903861
- See also: The Stanley Medical Research Institute (SMRI) is a nonprofit organization supporting research on the causes of, and treatments for, schizophrenia and bipolar disorder. This current study was supported by the SMRI. — http://www.stanleyresearch.org